CLINICAL TRIAL: NCT00073450
Title: An Open-Label Phase 2 Study of Lonafarnib in Patients With Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of Lonafarnib in Patients With Recurrent Squamous Cell Carcinoma of the Head and Neck (Study P02530)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P02530
Record Dates: First submitted 2003-11-20; First posted 2003-11-24 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma, Squamous Cell; Head and Neck Neoplasms
Keywords: Squamous Cell Carcinoma of the Head & Neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — 2-(2-oxo-2-((3,7,11-trimethyl-2,6,10-dodecatrienyl)oxy)aminoethyl)phosphonic acid, (2,2-dimethyl-1-oxopropoxy)methyl ester sodium

INTERVENTIONS:
Drug: Farnesyl Protein Transferase Inhibitor

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an oral Farnesyl Protein Transferase Inhibitor (Lonafarnib/SCH 6636) as a single agent in Adult Patients With Squamous Cell Carcinoma of the Head & Neck and will help determine if further development is justified.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head & neck.
* Age greater than or equal to 18.
* ECOG performance status of 0 to 1
* Measurable malignant disease.
* Patients that have failed at least one platinum-containing regimen and have received no more than three prior regimens and do not have other curative treatment options.
* Patients must be at least 2 wks post surgery or radiation therapy
* Patients must be at least 4 weeks post chemotherapy
* Meets protocol requirements for specified laboratory values.
* Written informed consent and cooperation of patient.
* Appropriate use of effective contraception if of childbearing potential.
* No investigational drugs of any type within 30 days prior to administration.

Exclusion Criteria:

* Prior exposure to farnesyl transferase inhibitors
* Medical conditions that would interfere with taking oral medications.
* Patients with significant QTc prolongation at baseline (>500 msec.)
* Pregnant or nursing women
* Known HIV positivity or AIDS-related illness.
* Concomitant chemotherapy, hormonal therapy, radiotherapy or immunotherapy
* Patients with any signs of involvement of the dura, meninges, or brain.
* Patients with squamous cell carcinoma of the nasopharynx
* Patients who currently have other cancers or have been treated in the last 5 years for any other malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-09; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

REFERENCES:
- [Result] Hanrahan EO, Kies MS, Glisson BS, Khuri FR, Feng L, Tran HT, Ginsberg LE, Truong MT, Hong WK, Kim ES. A phase II study of Lonafarnib (SCH66336) in patients with chemorefractory, advanced squamous cell carcinoma of the head and neck. Am J Clin Oncol. 2009 Jun;32(3):274-9. doi: 10.1097/COC.0b013e318187dd57. PMID 19433965